CLINICAL TRIAL: NCT07170865
Title: Assessment of the Dynamic Impact of Non-Invasive Ventilation on Diaphragmatic Ultrasound in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Dynamic Impact of NIV on Diaphragmatic Ultrasound in Patients With Amyotrophic Lateral Sclerosis
Acronym: EchoDia
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC25.0186
Record Dates: First submitted 2025-08-19; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-06

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS); Non Invasive Ventilation (NIV)
Keywords: Amyotrophic Lateral Sclerosis (ALS); Non invasive ventilation (NIV); Diaphragmatic ultrasound; diaphragmatic excursion; ultrasound; diaphragmatic thickening
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this pilot observational study is to learn about the dynamic impact of the non invasive ventilation on the diaphragm in patient with amyotrophic lateral sclerosis. The main question it aims to answer : can diaphragmatic ultrasound detect differences in diaphragmatic motion (diaphragmactic excursion and diaphragmatic thickening between spontaneous breathing and non-invasive ventilation ?

Participants will receive diaphragmatic ultrasound assessments both under spontaneous breathing and during non-invasive ventilation on their day hospital evaluation for ventilatory support.

DETAILED DESCRIPTION:
Each diaphragmatic ultrasound assessment will be performed on both the right and left hemidiaphragms, with the patient in a semi-recumbent position at 30°, during a maximal inspiratory effort. The following parameters will be measured:

* Diaphragmatic excursion using M-mode ultrasound with a low-frequency convex (abdominal) probe via a subcostal approach
* Diaphragmatic thickening using B-mode ultrasound with a high-frequency linear (vascular) probe via the lateral axillary line

Measurements will be obtained during spontaneous breathing and after 10 to 20 minutes of non-invasive ventilation (NIV), using ventilator settings deemed optimally adjusted by the supervising physician.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old)
* Diagnosis of bulbar or spinal amyotrophic lateral sclerosis (ALS) established by a neurologist
* Indication for non-invasive ventilation (NIV) confirmed by the referring pulmonologist for daytime and/or nocturnal alveolar hypoventilation

Exclusion Criteria:

* Continuous (24-hour) non-invasive ventilation
* Patient refusal to participate
* Individual under legal guardianship or judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of bulbar or spinal amyotrophic lateral sclerosis (ALS) established by a neurologist
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Composite : - Diaphragmatic excursion variation (DE) - Diaphragmatic thickening variation (DT) | Day 1
  Both DE and DT will be measured under spontaneous bretahing and under NIV. The outcomes will be compared, and the percentage variation between the two conditions will be recorded

SECONDARY OUTCOMES:
Changes in transcutaneous carbon dioxide (TcCO₂) levels | Day 1
  The variation in TcCO₂ will be measured and compared with the variations in DE and DT to determine whether there is a correlation.
NIV Tolerance | Day 1
  NIV tolerance will be assessed using a numerical subjective scale from 0 to 10. The tolerance numercial scale will then be compared with variations in DE and DT to determine whether there is a correlation.
Pathophysiological type of ALS | Day 1
  For each patient, the bulbar type or the spinal type of ALS will be recorded. Subgroups analyses between spinal ALS and bulbar ALS. Some differences are to be expected.
Adherence of NIV | Day 1
  If a NIV is already instaured, the average adherence in hours per 24 hours will be recorded
  - Subgroupes analyses between < 8 hours/24h NIV adherence, and 8 hours/24h or more NIV adherence

CONTACTS AND LOCATIONS:
Overall Officials: Christel Saint Raymond, Doctor, Study Director — CHU Grenoble Alpes
Locations (1):
- CHU Grenoble-Alpes, Grenoble, Isère, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Georges M, Perez T, Rabec C, Jacquin L, Finet-Monnier A, Ramos C, Patout M, Attali V, Amador M, Gonzalez-Bermejo J, Salachas F, Morelot-Panzini C. Proposals from a French expert panel for respiratory care in ALS patients. Respir Med Res. 2022 May;81:100901. doi: 10.1016/j.resmer.2022.100901. Epub 2022 Mar 3. PMID 35378353
- [Background] Kang HW, Kim TO, Lee BR, Yu JY, Chi SY, Ban HJ, Oh IJ, Kim KS, Kwon YS, Kim YI, Kim YC, Lim SC. Influence of diaphragmatic mobility on hypercapnia in patients with chronic obstructive pulmonary disease. J Korean Med Sci. 2011 Sep;26(9):1209-13. doi: 10.3346/jkms.2011.26.9.1209. Epub 2011 Sep 1. PMID 21935278
- [Background] Cammarota G, Sguazzotti I, Zanoni M, Messina A, Colombo D, Vignazia GL, Vetrugno L, Garofalo E, Bruni A, Navalesi P, Avanzi GC, Della Corte F, Volpicelli G, Vaschetto R. Diaphragmatic Ultrasound Assessment in Subjects With Acute Hypercapnic Respiratory Failure Admitted to the Emergency Department. Respir Care. 2019 Dec;64(12):1469-1477. doi: 10.4187/respcare.06803. Epub 2019 Aug 27. PMID 31455684
- [Background] Qian Z, Yang M, Li L, Chen Y. Ultrasound assessment of diaphragmatic dysfunction as a predictor of weaning outcome from mechanical ventilation: a systematic review and meta-analysis. BMJ Open. 2018 Oct 4;8(9):e021189. doi: 10.1136/bmjopen-2017-021189. PMID 30287605
- [Background] Marques MR, Pereira JM, Paiva JA, de Casasola-Sanchez GG, Tung-Chen Y. Ultrasonography to Access Diaphragm Dysfunction and Predict the Success of Mechanical Ventilation Weaning in Critical Care: A Narrative Review. J Ultrasound Med. 2024 Feb;43(2):223-236. doi: 10.1002/jum.16363. Epub 2023 Nov 2. PMID 37915259
- [Background] Pinto S, Alves P, Pimentel B, Swash M, de Carvalho M. Ultrasound for assessment of diaphragm in ALS. Clin Neurophysiol. 2016 Jan;127(1):892-897. doi: 10.1016/j.clinph.2015.03.024. Epub 2015 Apr 25. PMID 25971723
- [Background] Fantini R, Mandrioli J, Zona S, Antenora F, Iattoni A, Monelli M, Fini N, Tonelli R, Clini E, Marchioni A. Ultrasound assessment of diaphragmatic function in patients with amyotrophic lateral sclerosis. Respirology. 2016 Jul;21(5):932-8. doi: 10.1111/resp.12759. Epub 2016 Mar 19. PMID 26994409
- [Background] Bourke SC, Tomlinson M, Williams TL, Bullock RE, Shaw PJ, Gibson GJ. Effects of non-invasive ventilation on survival and quality of life in patients with amyotrophic lateral sclerosis: a randomised controlled trial. Lancet Neurol. 2006 Feb;5(2):140-7. doi: 10.1016/S1474-4422(05)70326-4. PMID 16426990
- [Background] Su WM, Cheng YF, Jiang Z, Duan QQ, Yang TM, Shang HF, Chen YP. Predictors of survival in patients with amyotrophic lateral sclerosis: A large meta-analysis. EBioMedicine. 2021 Dec;74:103732. doi: 10.1016/j.ebiom.2021.103732. Epub 2021 Dec 1. PMID 34864363
- [Background] Brown RH, Al-Chalabi A. Amyotrophic Lateral Sclerosis. N Engl J Med. 2017 Jul 13;377(2):162-172. doi: 10.1056/NEJMra1603471. No abstract available. PMID 28700839
- [Background] Lo Coco D, Marchese S, Pesco MC, La Bella V, Piccoli F, Lo Coco A. Noninvasive positive-pressure ventilation in ALS: predictors of tolerance and survival. Neurology. 2006 Sep 12;67(5):761-5. doi: 10.1212/01.wnl.0000227785.73714.64. Epub 2006 Aug 9. PMID 16899545
- [Background] Schenesse D, Mouillot P, Rabec C, Barnestein R, Tankere P, Giboulot M, Bonniaud P, Georges M. [Diaphragmatic ultrasonography for the pulmonologist: Technique and clinical use]. Rev Mal Respir. 2024 Jan;41(1):1-17. doi: 10.1016/j.rmr.2023.10.005. Epub 2023 Nov 18. French. PMID 37980184
- [Background] Boussuges A, Bregeon F, Blanc P, Gil JM, Poirette L. Characteristics of the paralysed diaphragm studied by M-mode ultrasonography. Clin Physiol Funct Imaging. 2019 Mar;39(2):143-149. doi: 10.1111/cpf.12549. Epub 2018 Oct 16. PMID 30325572
- [Background] Hiwatani Y, Sakata M, Miwa H. Ultrasonography of the diaphragm in amyotrophic lateral sclerosis: clinical significance in assessment of respiratory functions. Amyotroph Lateral Scler Frontotemporal Degener. 2013 Mar;14(2):127-31. doi: 10.3109/17482968.2012.729595. Epub 2012 Oct 30. PMID 23110443
- [Background] Fantini R, Tonelli R, Castaniere I, Tabbi L, Pellegrino MR, Cerri S, Livrieri F, Giaroni F, Monelli M, Ruggieri V, Fini N, Mandrioli J, Clini E, Marchioni A. Serial ultrasound assessment of diaphragmatic function and clinical outcome in patients with amyotrophic lateral sclerosis. BMC Pulm Med. 2019 Aug 27;19(1):160. doi: 10.1186/s12890-019-0924-5. PMID 31455341
- [Background] Spiliopoulos KC, Lykouras D, Veltsista D, Skaramagkas V, Karkoulias K, Tzouvelekis A, Chroni E. The utility of diaphragm ultrasound thickening indices for assessing respiratory decompensation in amyotrophic lateral sclerosis. Muscle Nerve. 2023 Nov;68(6):850-856. doi: 10.1002/mus.27980. Epub 2023 Oct 10. PMID 37814924
- [Background] Czaplinski A, Yen AA, Appel SH. Forced vital capacity (FVC) as an indicator of survival and disease progression in an ALS clinic population. J Neurol Neurosurg Psychiatry. 2006 Mar;77(3):390-2. doi: 10.1136/jnnp.2005.072660. PMID 16484652